CLINICAL TRIAL: NCT03384719
Title: The Effect of Milk Protein vs. Blends of Milk and Plant Protein on Growth Markers in 7-8 Year Old Healthy Danish Children
Brief Title: The Effect of Milk Protein vs Blends of Milk and Plant Protein on Growth Markers in 7-8 Year Old Healthy Danish Children
Acronym: PROGRO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Arla Foods (Industry); University of Aarhus (Other)
Responsible Party: Principal Investigator, Christian Mølgaard, Professor, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: D221
Record Dates: First submitted 2017-12-13; First posted 2017-12-27 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2017-12

CONDITIONS: Growth Acceleration; Growth; Stunting, Nutritional
Keywords: Growth factor; Protein; Milk protein; Plant protein; Insulin-like growth factor-1 (IGF-1); Insulin; Insulin-like growth factor-binding protein-3 (IGFBP-3)
MeSH Terms: conditions — Growth Disorders; Insulin Resistance | interventions — Proteins; Milk

STUDY DESIGN:
Intervention Model Description: The study is a randomized, controlled, double-blind, parallel food intervention study with 3 study arms
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 35 g protein (30% milk + 70% rapeseed) (Experimental): 35 g protein per day (30% milk + 70% rapeseed) provided as a powder to be consumed every morning and evening
  Interventions: Dietary Supplement: 35 g protein (30% milk + 70% rapeseed)
- 35 g protein (54% milk + 46% rapeseed) (Experimental): 35 g protein per day (54% milk + 46% rapeseed) provided as a powder to be consumed every morning and evening
  Interventions: Dietary Supplement: 35 g protein (54% milk + 46% rapeseed)
- 35 g protein (100% milk) (Active Comparator): 35 g protein per day (100% milk) provided as a powder to be consumed every morning and evening
  Interventions: Dietary Supplement: 35 g protein (100% milk)

INTERVENTIONS:
Dietary Supplement: 35 g protein (30% milk + 70% rapeseed) — The daily amount of 35 g of protein is provided as a powder. The powder is packed in two separate sachets to be consumed in the morning and evening. Each sachet contains approximately 60 g of powder. The powder is mixed with liquid before intake.
  Protein powder ingredients (all are food quality):
  * Milk protein: Skimmed milk powder (Arla Foods, Viby, Denmark)
  * Rapeseed protein isolate: Isolexx® (BioExx, Saskatoon, Canada)
  * Other ingredients: lactose, sucrose, flavors, artificial sweeteners. The protein powders for each treatment group are standardized to contain the same amount of energy and lactose per day.
  Arms: 35 g protein (30% milk + 70% rapeseed)
Dietary Supplement: 35 g protein (54% milk + 46% rapeseed) — The daily amount of 35 g of protein is provided as a powder. The powder is packed in two separate sachets to be consumed in the morning and evening. Each sachet contains approximately 60 g of powder. The powder is mixed with liquid before intake.
  Protein powder ingredients (all are food quality):
  * Milk protein: Skimmed milk powder (Arla Foods, Viby, Denmark)
  * Rapeseed protein isolate: Isolexx® (BioExx, Saskatoon, Canada)
  * Other ingredients: lactose, sucrose, flavors, artificial sweeteners. The protein powders for each treatment group are standardized to contain the same amount of energy and lactose per day.
  Arms: 35 g protein (54% milk + 46% rapeseed)
Dietary Supplement: 35 g protein (100% milk) — The daily amount of 35 g of protein is provided as a powder. The powder is packed in two separate sachets to be consumed in the morning and evening. Each sachet contains approximately 60 g of powder. The powder is mixed with liquid before intake.
  Protein powder ingredients (all are food quality):
  * Milk protein: Skimmed milk powder (Arla Foods, Viby, Denmark)
  * Other ingredients: lactose, sucrose, flavors, artificial sweeteners. The protein powders for each treatment group are standardized to contain the same amount of energy and lactose per day.
  Arms: 35 g protein (100% milk)

SUMMARY:
The purpose of PROGRO is to determine which combinations of milk and plant proteins are optimal to promote growth factors in children

DETAILED DESCRIPTION:
The main objective is to assess how different protein blends affect growth factors in children. There is evidence to support that milk protein increases growth in children in both high and low-income countries. Therefore milk protein is often used in food aid for undernourished children in low-income countries. The study investigates if plant protein can partially replace milk protein without affecting growth promotion negatively. Plant protein could potentially reduce food aid costs and at the same time be a more sustainable protein source.

The PROGRO study is a 3-arm randomized, controlled trial. The effect of consuming 35 g pure milk protein/day is compared to intake of 35 g milk and rapeseed protein/day (ratio 30:70 and 54:46, respectively) in 7-8 year old healthy Danish children. The intervention period is 4 weeks and measurements and blood sampling are performed at baseline, week 1 and week 4. A 3-day weighed dietary intake is recorded before each visit. The primary outcome is Insulin-like growth factor-1 (IGF-1).

ELIGIBILITY:
Inclusion Criteria:

* Age 7-8 years
* Healthy*
* The child is willing to consume protein powder twice a day for 4 weeks
* The child is not a picky eater and so does not mind trying new foods and flavours
* The child speaks Danish in order to understand the study procedures
* The parents read and speak Danish in order to be properly informed about the study procedures
* Written informed consent has been obtained

  * The principal investigator, who is blinded to study treatment, will perform a case-by-case medical evaluation of children with any signs of being unhealthy or having any illness or taking medication at the time of admission. If the conditions are considered to potentially affect protein metabolism or growth, the children will not be included. If a child is acutely ill at the scheduled time of study start, the child cannot be included. But the child may be included later when the acute illness has resolved

Exclusion Criteria:

* The child drinks more than 350 ml of milk per day
* Known or suspected allergy, sensitization or intolerance to milk (protein or lactose), rapeseed or mustard
* Any acute illness*
* Chronic illness or disease that may affect protein metabolism or growth*
* Chronic intake of medicine that may affect protein metabolism or growth*
* Concomitant participation in other studies involving dietary supplements or blood sampling
* Living in a household with another participating child

  * The principal investigator, who is blinded to study treatment, will perform a case-by-case medical evaluation of children with any signs of being unhealthy or having any illness or taking medication at the time of admission. If the conditions are considered to potentially affect protein metabolism or growth, the children will not be included. If a child is acutely ill at the scheduled time of study start, the child cannot be included. But the child may be included later when the acute illness has resolved

Ages: 7 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 129 (Actual)
Dates: Start 2018-01-18 (Actual); Primary Completion 2018-12-18 (Actual); Study Completion 2018-12-18 (Actual)

PRIMARY OUTCOMES:
Change in IGF-I between study arms | from baseline to week 4
  Blood sample

SECONDARY OUTCOMES:
Change in IGF-1 within study arms | from baseline to week 4
  Blood sample
Change in IGF-1 between and within study arms | from baseline to week 1
  Blood sample
Change in IGFBP-3 between and within study arms | from baseline to week 1 and week 4, respectively
  Blood sample
Change in the ratio IGF-1/IGFBP-3 between and within study arms | from baseline to week 1 and week 4, respectively
  Blood sample. Concentration of IGF-1 divided by the concentration of IGFBP-3.
Change in insulin between and within study arms | from baseline to week 1 and week 4, respectively
  Blood sample
Change in relative insulin resistance between and within study arms | from baseline to week 1 and week 4, respectively
  Blood sample
Change in beta cell function between and within study arms | from baseline to week 1 and week 4, respectively
  Blood sample
Change in beta cell function/insulin resistance between and within study arms | from baseline to week 1 and week 4, respectively
  Blood sample. Beta cell function divided by insulin resistance.

OTHER OUTCOMES:
Change in weight | from baseline to week 1 and week 4, respectively
  The weight is measured once on a digital weighing scale (Tanita MC 780) in kg
Change in body mass index (BMI) | from baseline to week 1 and week 4, respectively
  BMI = weight divided by height squared (kg/m2). Weight is measured once using a digital weighing scale while the child is wearing underwear (Tanita MC 780, unit: kg) and height is measured three times to the nearest millimeter using a stadiometer (unit: meter).
Change in waist circumference | from baseline to week 1 and week 4, respectively
  Measured three times to the nearest millimeter using a non-elastic measuring tape
Change in bio impedance | from baseline to week 1 and week 4, respectively
  Tanita MC 780MA segmental multi frequency body composition analyzer
Change in subscapular and triceps skinfolds | from baseline to week 1 and week 4, respectively
  Subscapular and triceps skinfolds are measured three times to the non-dominant side to the nearest 0.2 millimeter using a Harpenden skinfold caliper while the child is standing
Change in free amino acids in plasma | from baseline to week 1 and week 4, respectively
  Blood sample
Change in height | from baseline to week 1 and week 4, respectively
  Height is measured three times to the nearest millimeter using a stadiometer
Change in blood pressure | from baseline to week 1 and week 4, respectively
  Blood pressure will be measured three times by an automated medical device while the child is lying down. Blood pressure is measured after 10 minutes rest
Change in pulse rate | from baseline to week 1 and week 4, respectively
  Blood pressure and pulse will be measured three times by an automated medical device while the child is lying down. Blood pressure and pulse are measured after 10 minutes rest
Change in appetite hormones | from baseline to week 1 and week 4, respectively
  Blood sample: leptin
Change in appetite hormones | from baseline to week 1 and week 4, respectively
  Blood sample: adiponectin
Change in bone turnover marker: CTX (C-terminal telopeptide, carboxy-terminal collagen crosslinks) | from baseline to week 1 and week 4, respectively
  Blood sample
Change in bone specific alkaline phosphatase | from baseline to week 1 and week 4, respectively
  Blood sample
Change in osteocalcin | from baseline to week 1 and week 4, respectively
  Blood sample
Change in genetics | from baseline to week 1 and week 4, respectively
  Blood sample: epigenetics and genes related to the study outcomes (single nucleotides polymorphisms (SNPs) and genome wide association studies (GWAS), NOT full genome sequencing
Change in metabolomics related to the study outcomes | from baseline to week 1 and week 4, respectively
  Blood sample
Change in proteomics related to the study outcomes | from baseline to week 1 and week 4, respectively
  Blood sample

CONTACTS AND LOCATIONS:
Overall Officials: Christian Mølgaard, professor, Principal Investigator — University of Copenhagen; Benedikte Grenov, postdoc, Study Chair — University of Copenhagen; Anni Larnkjær, PhD, Study Chair — University of Copenhagen; Camilla T. Damsgaard, Associate Professor, Study Chair — University of Copenhagen
Locations (1):
- Department of Nutrition, Exercise and Sports, Copenhagen, Frederiksberg, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Grenov B, Larnkjaer A, Ritz C, Michaelsen KF, Damsgaard CT, Molgaard C. The effect of milk and rapeseed protein on growth factors in 7-8 year-old healthy children - A randomized controlled trial. Growth Horm IGF Res. 2021 Oct-Dec;60-61:101418. doi: 10.1016/j.ghir.2021.101418. Epub 2021 Jul 21. PMID 34333391